CLINICAL TRIAL: NCT06723288
Title: A Multicenter, Cross-sectional Study to Describe the Conjunctiva and Tenon's Capsule Status of Healthy Subjects and nAMD/DME Patients Followed in Clinical Practice in Spain
Brief Title: A Study Conducted to Evaluate the Conjunctiva and Tenon's Capsule Status of Healthy Subjects and in Participants With Neovascular Age-related Macular Degeneration (nAMD)/Diabetic Macular Edema (DME)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MR45734
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: nAMD/DME Participants: Participants with nAMD/DME will be enrolled in this cohort given, they meet the eligibility criteria. The SD-OCT test will be conducted for all participants in this cohort. Additionally, swept source optical coherence tomography (SS-OCT) will be performed on the first 50 participants.
- Cohort B: Healthy Subjects: Healthy subjects who meet the eligibility criteria will be enrolled in this cohort. The SD-OCT test will be conducted for all subjects in this cohort. Additionally, SS-OCT will be performed on the first 50 healthy subjects.

SUMMARY:
The purpose of this study is to obtain conjunctiva and tenon's capsule thickness measurements in vivo using spectral domain-optical coherence tomography (SD-OCT) in participants with nAMD/DME and age-matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

For nAMD/DME participants:

- Diagnosis of nAMD/DME

For healthy subjects:

- Normal visual function

Exclusion Criteria:

* Current or past treatment for glaucoma (only for healthy subjects)
* Dry eye disease except those treated only with artificial tears
* Ocular hypertension treated with hypotensive drugs
* Pterygium
* Strabismus
* Previous ocular surgery except cataract surgery
* Cataract surgery with scleral incision
* Current contact lens wearers
* Myopia with more than 6 diopters
* Corneal transplant
* History of ocular surface inflammation
* Active or recent conjunctivitis infection
* Pregnancy
* Participant who has already received an IVT injection in the superotemporal quadrant (only for nAMD/DME participants)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with nAMD or DME and age-matched healthy subjects from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 736 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Cohorts A and B: Conjunctival Epithelium Thickness Measured Using SD-OCT | At study visit (Day 1)
Cohorts A and B: Conjunctival Stroma Thickness Measured Using SD-OCT | At study visit (Day 1)
Cohorts A and B: Tenon's Capsule Thickness Measured Using SD-OCT | At study visit (Day 1)
Cohorts A and B: Sum of Conjunctival Epithelium Thickness, Conjunctival stroma and Tenon's Capsule Measured Using SD-OCT | At study visit (Day 1)
Cohorts A and B: Number of Participants in Age Groups 45-54, 55-64, 65-74, >=75 | At study visit (Day 1)

SECONDARY OUTCOMES:
Cohort A: Previous Intravitreal (IVT) Injections (Yes/No) | At study visit (Day 1)
Cohorts A and B: Conjunctival Epithelium Thickness Measured Using SS-OCT | At study visit (Day 1)
Cohorts A and B: Conjunctival Stroma Thickness Measured Using SS-OCT | At study visit (Day 1)
Cohorts A and B: Tenon's Capsule Thickness Measured Using SS-OCT | At study visit (Day 1)
Cohorts A and B: Sum of Conjunctival Epithelium Thickness, Conjunctival stroma and Tenon's Capsule Measured Using SS-OCT | At study visit (Day 1)
Cohorts A and B: Scleral Thickness Measured Using SS-OCT | At study visit (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Spain (20):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Oftalvist Valencia, Burjassot, Valencia
  - Centro de Oftalmologia Barraquer, Barcelona
  - Institut de la Macula i la retina, Barcelona
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Arruzafa. Servicio de Oftalmologia, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Clinica Baviera, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Virgen del Rocio, Seville
  - Clinica Oftalmologica Aiken, Valencia
  - Hospital Arnau de Vilanova (Valencia), Valencia
  - Hospital Universitario Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No